CLINICAL TRIAL: NCT03189745
Title: A PHASE IIIB, OPEN STUDY TO EVALUATE THE IMMUNOGENICITY, REACTOGENICITY AND SAFETY OF A BOOSTER DOSE OF MENACWY-TT VACCINE ADMINISTERED 10 YEARS AFTER HEALTHY SUBJECTS AGED 11-17 YEARS RECEIVED EITHER MENACWY-TT VACCINE (NIMENRIX(REGISTERED)) OR MENCEVAX ACWY(REGISTERED).
Brief Title: A Study To Evaluate A Booster Dose Of Menacwy-tt Vaccine Administered 10 Years After Healthy Subjects Aged 11-17 Years Received Either Menacwy-tt Vaccine (Nimenrix(Registered)) Or Mencevax Acwy(Registered).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MENACWY-TT-101; C0921005 (Other: Alias Study Number); 2013-001512-29 (EudraCT Number); 116724 (Other: Alias Study Number)
Record Dates: First submitted 2017-05-23; First posted 2017-06-16 (Actual); Results first posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-09

CONDITIONS: Meningococcal ACWY Disease
MeSH Terms: interventions — tetravalent meningococcal serogroups A, C, W-135 and Y tetanus toxoid conjugate vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MenACWY-TT Booster (Experimental): 10 year booster dose of MenACWY
  Interventions: Biological: MenACWY-TT

INTERVENTIONS:
Biological: MenACWY-TT — Single dose of MenACWY-TT given 10 years after first vaccine with either MenACWY-TT or Mencevax ACWY

SUMMARY:
This study will evaluate the immunogenicity, reactogenicity and safety of a booster dose of MenACWY-TT vaccine administered 10 years after healthy subjects aged 11-17 years received either MenACWY-TT vaccine (Nimenrix) or Mencevax ACWY

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply, with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits).
* Written informed consent obtained from the subject prior to performing any study specific procedure.
* Healthy male or female subjects as established by medical history and history-directed physical examination before entering into the study.
* Having completed the vaccination in study MenACWY-TT-036 (109069) as per protocol.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Non-childbearing potential is defined as pre-menarche, hysterectomy, bilateral ovariectomy or post-menopause.

Please refer to the GLOSSARY OF TERMS for the definitions of menarche and post-menopause.

* Male subjects able to father children and female subjects of childbearing potential (including females who have had tubal ligation) and at risk for pregnancy may be enrolled in the study, if the subject:
* has practiced adequate contraception for 30 days prior to vaccination, and
* has a negative pregnancy test on the day of vaccination (for females only), and
* has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose. For corticosteroids, this will be 10 mg/day prednisone, or equivalent. Inhaled, topical, and intra-articular steroids are allowed.
* Administration of a vaccine not foreseen by the study protocol within the period starting 30 days before and ending 30 days after the study vaccine dose, with the exception of a licensed inactivated influenza vaccine which can be administered at any time during the study according to the local recommendations.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the study vaccination or planned administration during the booster vaccination phase of the study (i.e. between Visit 1 and Visit 2).
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Previous vaccination with meningococcal vaccine except the meningococcal vaccination received in the MenACWY-TT-036 study.
* Any confirmed or suspected immunosuppressive or immunodeficient condition (congenital or secondary), including human immunodeficiency virus infection, based on medical history and physical examination (no laboratory testing required).
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine, and history of serious allergic reaction (anaphylaxis) following the administration of vaccine(s).
* Major congenital defects or serious chronic illness.
* History of any neurological disorders or seizures, including GBS. History of a simple, single febrile seizure is permitted.
* Acute disease and/or fever at the time of vaccination.
* Fever is defined as temperature ≥ 37.5°C for oral, axillary or tympanic route, or ≥ 38.0°C for rectal route. The preferred route for recording temperature in this study will be oral.
* Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be vaccinated at the discretion of the investigator.
* Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees directly involved in the conduct of the study.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Male subjects able to father children who are planning to discontinue contraceptive precautions.

Ages: 20 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 229 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Research Institute for Tropical Medicine, Muntinlupa City, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=MENACWY-TT-101

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who received either MenACWY-TT (NIMENRIX) or Mencevax ACWY vaccine in study 109069 (NCT00464815) were administered a MenACWY-TT booster vaccination in this study and evaluated for immunogenicity, reactogenicity and safety parameters.
Groups:
- ACWY-TT Group: Participants received a single 0.5 milliliter (mL) dose of meningococcal serogroups A, C, W-135, Y tetanus toxoid conjugate (MenACWY-TT) vaccine intramuscularly as primary vaccination in study 109069 (NCT00464815) and then 10 years post primary vaccination received a single 0.5 mL dose of MenACWY-TT vaccine intramuscularly as booster vaccination. Participants were also evaluated for long-term persistence (of immune response and safety) at year 10 post primary vaccination.
- MenPS Group: Participants received a single 0.5 mL dose of MencevaxACWY vaccine intramuscularly as primary vaccination in study 109069 (NCT00464815) and then 10 years post primary vaccination received a single 0.5 mL dose of MenACWY-TT vaccine intramuscularly as booster vaccination. Participants were also evaluated for long-term persistence (of immune response and safety) at year 10 post primary vaccination.
Period: Overall Study
Arm/Group | ACWY-TT Group | MenPS Group
Started | 170 | 59
Completed | 169 | 58
Not Completed | 1 | 1
Not completed — Conflict in work schedule of participant | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants enrolled in the study.
Groups:
- ACWY-TT Group: Participants received a single 0.5 mL dose of MenACWY-TT vaccine intramuscularly as primary vaccination in study 109069 (NCT00464815) and then 10 years post primary vaccination received a single 0.5 mL dose of MenACWY-TT vaccine intramuscularly as booster vaccination. Participants were also evaluated for long-term persistence (of immune response and safety) at year 10 post primary vaccination.
- Total: Total of all reporting groups
Arm/Group | ACWY-TT Group | MenPS Group | Total
Number analyzed (Participants) | 170 | 59 | 229
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.2 (1.9) | 24.0 (2.0) | 24.1 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 23 | 103
  Male | 90 | 36 | 126
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - South East Asian heritage | 170 | 59 | 229

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Booster Response in Terms of Serum Bactericidal Assay Using Rabbit Complement (rSBA) Titer Levels at 1 Month After Booster Vaccination
Description: Serogroups included: Neisseria meningitidis serogroup A (MenA), Neisseria meningitidis serogroup C (MenC), Neisseria meningitidis serogroup W-135 (MenW-135) and Neisseria meningitidis serogroup Y (MenY). The rSBA titer levels greater than or equal to (>=) 1:32 for initially seronegative participants and at least four-fold increase in rSBA titer levels for initially seropositive participants, 1 month after booster vaccination were defined as booster response to meningococcal antigens and reported in this outcome measure. Initially seronegative participants were defined as participants with pre-vaccination rSBA titer levels below 1:8 and initially seropositive participants were defined as participants with pre-vaccination rSBA titer >=1:8. Data reported below is including both seropositive and seronegative participants.
Time Frame: 1 month after booster vaccination
Population: Booster according-to-protocol(ATP)Cohort for immunogenicity: met booster ATP cohort for safety, comply procedures in protocol, meeting visit interval from primary vaccination(vac) in 109069 to booster vac,blood sampling intervals, had assay results with no vac before post booster vac blood draw.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 162 | 51
percentage of participants
  rSBA-MenA | 81.5 [74.6 to 87.1] | 84.3 [71.4 to 93.0]
  rSBA-MenC | 88.3 [82.3 to 92.8] | 66.7 [52.1 to 79.2]
  rSBA-MenW-135 | 95.7 [91.3 to 98.2] | 94.1 [83.8 to 98.8]
  rSBA-MenY | 87.0 [80.9 to 91.8] | 90.2 [78.6 to 96.7]

2. Secondary Outcome: Percentage of Participants With rSBA Titer Levels >=1:8 and >=1:128 for Each of the 4 Serogroups Before Booster Vaccination and 1 Month After Booster Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: Before booster vaccination, 1 month after booster vaccination (Vac)
Population: Booster ATP Cohort for immunogenicity: met requirements of booster ATP cohort for safety, comply procedures in protocol included meeting visit interval from primary vaccination in 109069(NCT00464815) to booster vaccination and blood sampling intervals, had assay results with no vaccine administered before post booster vaccination blood draw.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 162 | 51
percentage of participants
  rSBA-MenA: >=1:8; Before booster vaccination | 85.2 [78.8 to 90.3] | 80.4 [66.9 to 90.2]
  rSBA-MenA: >=1:8;1 month after booster vaccination | 100.0 [97.7 to 100.0] | 100.0 [93.0 to 100.0]
  rSBA-MenC: >=1:8; Before booster vaccination | 90.1 [84.5 to 94.2] | 82.4 [69.1 to 91.6]
  rSBA-MenC: >=1:8;1 month after booster vaccination | 100.0 [97.7 to 100.0] | 100.0 [93.0 to 100.0]
  rSBA-MenW-135: >=1:8; Before booster vaccination | 71.6 [64.0 to 78.4] | 43.1 [29.3 to 57.8]
  rSBA-MenW-135:>=1:8;1month after booster vac | 100.0 [97.7 to 100.0] | 100.0 [93.0 to 100.0]
  rSBA-MenY: >=1:8; Before booster vaccination | 90.7 [85.2 to 94.7] | 49.0 [34.8 to 63.4]
  rSBA-MenY: >=1:8;1 month after booster vaccination | 100.0 [97.7 to 100.0] | 98.0 [89.6 to 100.0]
  rSBA-MenA: >=1:28; Before booster vaccination | 81.5 [74.6 to 87.1] | 76.5 [62.5 to 87.2]
  rSBA-MenA:>=1:28;1 month after booster vaccination | 100.0 [97.7 to 100.0] | 100.0 [93.0 to 100.0]
  rSBA-MenC: >=1:28; Before booster vaccination | 77.2 [69.9 to 83.4] | 62.7 [48.1 to 75.9]
  rSBA-MenC:>=1:28;1 month after booster vaccination | 100.0 [97.7 to 100.0] | 100.0 [93.0 to 100.0]
  rSBA-MenW-135: >=1:28; Before booster vaccination | 64.8 [56.9 to 72.1] | 25.5 [14.3 to 39.6]
  rSBA-MenW-135:>=1:28;1month after booster vac | 100.0 [97.7 to 100.0] | 98.0 [89.6 to 100.0]
  rSBA-MenY: >=1:28; Before booster vaccination | 85.2 [78.8 to 90.3] | 39.2 [25.8 to 53.9]
  rSBA-MenY:>=1:28;1 month after booster vaccination | 100.0 [97.7 to 100.0] | 96.1 [86.5 to 99.5]

3. Secondary Outcome: rSBA Geometric Mean Titers for Each of the 4 Serogroups Before Booster Vaccination and 1 Month After Booster Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY. rSBA titers were expressed as the reciprocal of the highest serum last dilution resulting in at least 50 percentage (%) reduction of meningococcal colony-forming units.
Time Frame: Before booster vaccination, 1 month after booster vaccination
Population: Booster ATP Cohort for immunogenicity: met requirements of booster ATP cohort for safety, comply procedures in protocol included meeting visit interval from primary vaccination in 109069 (NCT00464815) to booster vaccination and blood sampling intervals, had assay results with no vaccine administered before post booster vaccination blood draw.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 162 | 51
titers
  rSBA-MenA; Before booster vaccination | 248.4 [181.4 to 340.2] | 142.7 [80.5 to 252.9]
  rSBA-MenA;1 month after booster vaccination | 3760.1 [3268.3 to 4325.9] | 2956.0 [2040.5 to 4282.1]
  rSBA-MenC; Before booster vaccination | 244.2 [181.6 to 328.5] | 177.4 [86.1 to 365.3]
  rSBA-MenC;1 month after booster vaccination | 8697.7 [7391.2 to 10235.1] | 3879.3 [2714.6 to 5543.7]
  rSBA-MenW-135; Before booster vaccination | 145.5 [97.6 to 217.1] | 16.4 [9.2 to 29.4]
  rSBA-MenW-135;1 month after booster vaccination | 11243.4 [9366.8 to 13496.0] | 3674.0 [2353.9 to 5734.4]
  rSBA-MenY; Before booster vaccination | 446.5 [332.7 to 599.1] | 32.9 [17.1 to 63.3]
  rSBA-MenY; 1 month after booster vaccination | 7584.8 [6748.4 to 8524.7] | 3295.5 [1998.7 to 5433.7]

4. Secondary Outcome: Percentage of Participants With Anti-Tetanus Toxoid (Anti-TT) Concentrations >=0.1 International Units Per Millilitre (IU/mL), >=1.0 IU/mL Before Booster Vaccination and 1 Month After Booster Vaccination
Description: Tetanus toxoid (TT) was used as carrier in tetravalent meningococcal ACWY conjugate vaccine. Percentage of participants with anti-TT concentration >=0.1 IU/mL, >=1.0 IU/mL were summarized.
Time Frame: Before booster vaccination, 1 month after booster vaccination
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 162 | 51
percentage of participants
  >=0.1 IU/mL; Before booster vaccination | 86.4 [80.2 to 91.3] | 54.9 [40.3 to 68.9]
  >=0.1 IU/mL;1 month after booster vaccination | 98.8 [95.6 to 99.9] | 96.1 [86.5 to 99.5]
  >=1.0 IU/mL; Before booster vaccination | 38.3 [30.8 to 46.2] | 27.5 [15.9 to 41.7]
  >=1.0 IU/mL; 1 month after booster vaccination | 92.0 [86.7 to 95.7] | 82.4 [69.1 to 91.6]

5. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Anti-Tetanus Toxoid Before Booster Vaccination and 1 Month After Booster Vaccination
Description: TT was used as carrier in tetravalent meningococcal ACWY conjugate vaccine. The GMCs calculations was performed by taking the anti-log of the mean of the log concentration transformations. Antibody (Anti-TT) concentrations below the cut-off value (0.1 IU/mL) of the assay was given an arbitrary value of half the cut-off value for the purpose of GMC calculation.
Time Frame: Before booster vaccination, 1 month after booster vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 162 | 51
IU/mL
  Before booster vaccination | 0.608 [0.476 to 0.775] | 0.252 [0.154 to 0.411]
  1 month after booster vaccination | 5.057 [4.274 to 5.984] | 5.115 [3.073 to 8.514]

6. Secondary Outcome: Percentage of Participants With Solicited Local and General Adverse Events Within 4 Days After Booster Vaccination
Description: Solicited local reactions included pain, redness and swelling. Pain graded as: (0= none, 1= mild, not interfered/prevented normal activity, 2= moderate, painful when limb moved/interfered with normal activity, 3= severe, significant pain at rest/ prevented normal activity). Redness and swelling scored as:0= None, 1= 0 to less than or equal to (<=) 20 millimeter (mm), 2= greater than (>) 20 to <=50 mm, 3=>50 mm. Solicited general reactions: headache, fatigue, gastrointestinal (GI) events (nausea, vomiting, diarrhea /abdominal pain) graded as (0= normal, 1=mild/easily tolerated, 2=moderate/interfered with normal activity, 3=severe / prevented normal activity). Fever categorized as: 0= less than (<) 37.5 degree Celsius (C), 1= >=37.5 to <=38.5 degree C, 2= >38.5 to <=39.5 degree C, and 3= >39.5 degree C.
Time Frame: Within 4 days post booster vaccination (Day 0 to Day 3)
Population: Booster total vaccinated cohort (TVC) for safety included all vaccinated participants in study 109069 (NCT00464815) with a MenACWY-TT booster vaccine administration documented in study MENACWY-TT-101. Here, "Overall Number of Participants Analyzed" (N) signifies number of participants evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 169 | 58
percentage of participants
  Pain: Grade 1 | 29.0 | 31.0
  Pain: Grade 2 | 4.7 | 1.7
  Pain: Grade 3 | 1.2 | 0.0
  Redness: Grade 1 | 10.1 | 8.6
  Redness: Grade 2 | 0.0 | 0.0
  Redness: Grade 3 | 0.0 | 0.0
  Swelling: Grade 1 | 7.7 | 3.4
  Swelling: Grade 2 | 0.0 | 0.0
  Swelling: Grade 3 | 0.0 | 0.0
  Fatigue: Grade 1 | 16.0 | 19.0
  Fatigue: Grade 2 | 1.8 | 5.2
  Fatigue: Grade 3 | 0.0 | 0.0
  Fever: Grade 1 | 4.1 | 3.4
  Fever: Grade 2 | 0.0 | 0.0
  Fever: Grade 3 | 0.0 | 0.0
  GI: Grade 1 | 9.5 | 6.9
  GI: Grade 2 | 1.8 | 3.4
  GI: Grade 3 | 0.0 | 0.0
  Headache: Grade 1 | 21.3 | 15.5
  Headache: Grade 2 | 3.6 | 6.9
  Headache: Grade 3 | 0.6 | 0.0

7. Secondary Outcome: Percentage of Participants With Unsolicited Adverse Events (AEs) Within 31 Days After Booster Vaccination
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. And any AE reported in addition to those solicited during the clinical study. Also any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
Time Frame: 31 days after booster vaccination (Day 0 to Day 30)
Population: Booster TVC for safety included all vaccinated participants in study 109069 (NCT00464815) with a MenACWY-TT booster vaccine administration documented in study MENACWY-TT-101.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 170 | 59
percentage of participants | 9.4 [5.5 to 14.8] | 15.3 [7.2 to 27.0]

8. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs), Guillain-Barre Syndrome (GBS) and New Onset of Chronic Illnesses (NOCI) Within 31 Days After Booster Vaccination
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. GBS is a rare neurological disorder in which the body's immune system mistakenly attacks part of its peripheral nervous system-the network of nerves located outside of the brain and spinal cord. GBS can range from a very mild case with brief weakness to nearly devastating paralysis, leaving the person unable to breathe independently. All occurrences of GBS has to be reported as an SAE. New onset chronic illness included autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: Within 31 days after booster vaccination (Day 0 to Day 30)
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 170 | 59
percentage of participants
  SAEs | 0 | 0
  GBS | 0 | 0
  NOCI | 0 | 0

9. Secondary Outcome: Percentage of Participants With SAEs Related to Primary Vaccination and Any Events Related to Lack of Vaccine Efficacy After 10 Years of Primary Vaccination
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Occurrence of SAEs related to primary vaccination and any event related to lack of vaccine efficacy (i.e. meningococcal disease) from the participant's last visit in the primary study 109069 (NCT00464815) or in persistence study 112148 (NCT00974363); extension study: 109069 (NCT00464815) at Year 2, 3, 4, 5 after primary vaccination until entry in study MenACWYTT-101, which is extension of study 109069 (NCT00464815), 10 years post primary vaccination.
Time Frame: 10 years after primary vaccination
Population: The total cohort at Month 120 (10 years post primary vaccination) included all vaccinated participants from the vaccination of Study 109069 (NCT00464815) who return for the Month 120 follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 170 | 59
percentage of participants
  SAEs | 0 | 0
  Events related to lack of vac efficacy | 0 | 0

10. Other Pre Specified Outcome: Percentage of Participants With rSBA Titer Levels >=1:8 and >=1:128 For Each of the 4 Serogroups at 10 Years After Primary Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: 10 years after primary vaccination
Population: ATP Cohort for Persistence at Month 120: participants who eligible in Study 109069 (NCT00464815), received primary vaccination with MenACWY-TT or Mencevax ACWY during Study 109069, had assay results for at least one tested antigen at Month 120, did not received a meningococcal vaccine not planned in Study 109069 before Month 120 visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 163 | 53
percentage of participants
  rSBA-MenA: >=1:8 | 84.7 [78.2 to 89.8] | 81.1 [68.0 to 90.6]
  rSBA-MenC: >=1:8 | 90.2 [84.5 to 94.3] | 83.0 [70.2 to 91.9]
  rSBA-MenW-135: >=1:8 | 71.8 [64.2 to 78.5] | 41.5 [28.1 to 55.9]
  rSBA-MenY: >=1:8 | 90.8 [85.3 to 94.8] | 49.1 [35.1 to 63.2]
  rSBA-MenA: >=1:128 | 81.0 [74.1 to 86.7] | 77.4 [63.8 to 87.7]
  rSBA-MenC: >=1:128 | 77.3 [70.1 to 83.5] | 64.2 [49.8 to 76.9]
  rSBA-MenW-135: >=1:128 | 65.0 [57.2 to 72.3] | 24.5 [13.8 to 38.3]
  rSBA-MenY: >=1:128 | 85.3 [78.9 to 90.3] | 37.7 [24.8 to 52.1]

11. Other Pre Specified Outcome: Geometric Mean Titers With rSBA For Each of the 4 Serogroups at 10 Years After Primary Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY. rSBA titers were expressed as the reciprocal of the highest serum last dilution resulting in at least 50% reduction of meningococcal colony-forming units.
Time Frame: 10 years after primary vaccination
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | ACWY-TT Group | MenPS Group
Number analyzed (Participants) | 163 | 53
titers
  rSBA-MenA | 242.2 [176.6 to 332.3] | 153.7 [87.8 to 269.0]
  rSBA-MenC | 243.3 [181.1 to 326.7] | 182.2 [90.9 to 365.3]
  rSBA-MenW-135 | 146.0 [98.2 to 217.3] | 15.6 [8.9 to 27.4]
  rSBA-MenY | 446.9 [333.6 to 598.5] | 31.6 [16.8 to 59.6]

ADVERSE EVENTS:
Time Frame: Up to 31 days after booster vaccination (From Day 0 to Day 30). Solicited local and general reactions: Recorded by participants in e-diary within 4 days post booster vaccination (Day 0 to Day 3)
Description: All participants who received vaccine MenACWY-TT or Mencevax ACWY in study 109069 (NCT00464815) and received a MenACWY-TT booster dose in this study.
Arm/Group | ACWY-TT Group | MenPS Group
All-Cause Mortality (participants affected / at risk) | 0/170 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/170 | 0/59
Other Adverse Events (participants affected / at risk) | 83/170 | 30/59
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACWY-TT Group (N=170) | MenPS Group (N=59)
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal (Gastrointestinal disorders) | 19 | 6
Toothache (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 30 | 14
Injection site erythema (redness) (General disorders) | 17 | 5
Injection site pain (pain at injection site) (General disorders) | 59 | 19
Injection site swelling (swelling) (General disorders) | 13 | 2
Gastroenteritis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Pyuria (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Headache (Nervous system disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (3):
  • Study Protocol (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT03189745/Prot_000.pdf
  • Study Protocol (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT03189745/Prot_001.pdf
  • Statistical Analysis Plan (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/45/NCT03189745/SAP_002.pdf